CLINICAL TRIAL: NCT00662415
Title: Study Using Functional MRI to Examine Changes in the Brain in Unilateral Lower Limb Amputees Treated With Mirror Therapy for Phantom Limb Pain.
Brief Title: Examining Brain Changes Using Functional Magnetic Resonance Imaging (fMRI) in Amputees With Phantom Limb Pain Following Mirror Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: United States Department of Defense (U.S. Federal Agency)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Organization: Walter Reed Army Medical Center (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DCI-0771043
Record Dates: First submitted 2008-03-14; First posted 2008-04-21 (Estimated); Last update posted 2008-04-21 (Estimated); Status verified 2008-04

CONDITIONS: Phantom Limb Pain
Keywords: phantom limb pain; fMRI; mirror therapy
MeSH Terms: conditions — Phantom Limb | interventions — Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): 12 non-amputee control subjects will be scanned at 0, 2 and 4 weeks but will not recieve mirror therapy.
  Interventions: Behavioral: observation
- 2 (Experimental): 24 unilateral lower extremity amputee subjects will recieve daily mirror therapy for phantom limb pain and will be scanned at 0, 2, and 4 weeks.
  Interventions: Device: mirror-box treatment

INTERVENTIONS:
Device: mirror-box treatment — 15 minutes daily for 4 weeks
  Arms: 2
Behavioral: observation — observation
  Arms: 1

SUMMARY:
Almost everyone who has a traumatic limb amputated will experience a phantom limb - the vivid impression that the limb not only still is present, but also in many cases, painful. Preliminary data from study WRAMC WU# 05-71034, "Pilot study to assess the efficacy of mirror-box and mental visualization treatments on phantom limb pain" demonstrates that 4 weeks of mirror therapy is effective for treating phantom limb pain (PLP) and suggests that vision is a key component modulating PLP and may be the explanation for the efficacy of mirror therapy, as subjects view the reflected image of their intact limb while attempting to move the amputated, or phantom, limb. We propose conducting a study using functional magnetic resonance imaging (fMRI) to identify brain regions critical for the mirror effect and to study the relationship of visual activation to the sensation of phantom pain. Subjects will have an fMRI scan prior to starting therapy, 2 weeks after starting mirror therapy and again after 4 weeks of mirror therapy. Data will be gathered daily on the number of episodes of phantom limb pain, the average length of episodes, and the average intensity of pain.

DETAILED DESCRIPTION:
This is a prospective trial that will use fMRI to identify brain regions critical to the generation of PLP, examine the role of mirror therapy and the visual system in the de-activation of pain pathways, and observe how changes in the brain may be correlated with the level of PLP. Subjects must have PLP and have sustained a unilateral lower extremity amputation prior to enrollment. All subjects will be screened initially by a neurologist, physiatrist, or research coordinator according to the inclusion and exclusion criteria. A detailed medical history will be taken and documented, and a neurologist will conduct a documented physical examination. Subjects who do not meet the study inclusion criteria will not be eligible to participate in this research study, but will continue to receive current best practice of care. If a subject's pain becomes severe during the course of the study, pain medication will be available to them.

All subjects willing to participate in the study will be required to sign a DA 5303-R (see appendix for Voluntary Agreement Affidavit) prior to enrollment in the study. Once enrolled, all subjects will undergo baseline entry evaluations quantifying their current pain perception using the following evaluation tools: the Visual Analogue Scale (VAS) and the short version of the McGill Pain Questionnaire (Appendix 1) along with a short questionnaire on phantom limb pain frequency and duration (Appendix 5). Subjects will also be queried about their use of current pain medications along with the dosages on a weekly basis. Although helpful tools in the standard of care, the questionnaires completed by the subjects and the list of medications reported by the subjects in this study are for research data collection purposes only. In order to maintain subject confidentiality, only the subject's identification code-and not the subject's name-will appear on the questionnaires and evaluation forms. Subjects will be identified only through the use of coded identifiers. For instance, amputees would be coded as RLE1, RLE2, LLE1, LLE2, etc.

Dr. Jack Tsao, Katie Hughes, and Lindsay Hussey-Andersen will administer both the treatments and the questionnaires. They will train all research subjects on the appropriate technique for using a 2' X 4' mirror and perform the cognitive tests. Unilateral limb amputee subjects will be asked to place their intact foot in front of a mirror and then to view the mirror image of the intact foot moving while performing a series of foot movements with the amputated, or phantom, foot. The sequence of foot movements include: abduction of the great toe, adduction of the great toe, flexion of the foot, extension of the foot, inversion of the foot, eversion of the foot, rotation of the foot, flexion of the toes, and extension of the toes. These sessions will be supervised by a clinician or research coordinator and will occur 5 times a week for 4 weeks (20 days), with each session lasting 15 minutes. Prior to each daily treatment period, subjects will be asked to report PLP using the VAS and McGill forms and also to report the number and duration of PLP in the previous 24 hours. All subjects will also participate in rehabilitation therapy (muscle-strengthening exercises, use of prosthesis, and range of motion exercises) per standard medical care for limb amputation.

Concurrent use of pain medications and muscle relaxants is permitted and will be recorded by the research assistant in a medication diary (Appendix 2). Scores on the VAS and McGill pain questionnaire will be used to assess the subject's level of disability and to evaluate outcomes. Subjects will be evaluated weekly in the hospital for quantification of the amount of analgesic medications used (NSAIDs, muscle relaxants, opioids), and VAS and McGill scores will be quantified daily for 4 weeks. The primary outcome will be changes in brain areas which are activated at weeks 2 and 4 compared to areas activated prior to starting mirror therapy. Secondary outcomes will be pain relief on the VAS, with responders defined as subjects with a significant decrease in the VAS score. All respondents will be released from the study after the final pain evaluation at 4 weeks.

A research assistant will provide transportation to and from the National Institutes of Health (NIH) where the fMRI scans will take place. Amputee subjects will be asked to first use mental visualization to move their phantom foot and report their pain level, followed by viewing of their intact foot moving in a mirror while moving their phantom foot. fMRI scanning will be performed during both types of phantom foot movements to determine which additional brain regions are activated with visual observation. A fMRI will be done at the beginning of the study to establish a baseline and follow-up scanning will occur 2 and 4 weeks after daily mirror therapy begins to assess changes in brain activation. Fourteen (14) control subjects will be recruited and asked to perform the same tasks during the fMRI scans but will not undergo mirror therapy. Control subjects will complete the McGill pain questionnaire as well as the VAS during each of their 3 visits to NIH for fMRI scanning. All subjects will be queried about their current medication use on a weekly basis. Both amputee and control subjects will be a part of this study for one month; both will undergo 3 fMRI scanning sessions, interspersed by the same 2 week period. fMRI evaluations will take up to two (2) hours per session and mirror therapy will last fifteen (15) minutes, totaling six (6) hours of fMRI and five (5) hours and fifteen (15) minutes of mirror therapy.

ELIGIBILITY:
Inclusion Criteria:

For Amputee Subjects:

* Male or female subjects
* 18 to 75 years of age
* Active duty military
* Military healthcare beneficiary
* Military retiree
* Written informed consent and written authorization for use or release of health and research study information
* Unilateral lower limb amputation
* Right-handed
* Any level of prosthetic experience
* No prior history of vertebral disk disease/condition
* Sciatica
* Radiculopathy
* Neurological examination that will not interfere with participation in the study
* Minimum of 3 phantom limb pain episodes each week
* Degree of pain evaluated by VAS scoring a minimum of 3 cm at time of screening for entry into study.
* Ability to follow study instructions and likely to complete all required visits

For Control Subjects:

* Male or female subjects
* 18 to 75 years of age
* Written informed consent and written authorization for use or release of health and research study information
* Right-handed.
* No prior history of vertebral disk disease/condition
* Sciatica
* Radiculopathy
* Normal neurological examination
* Ability to follow study instructions and likely to complete all required visits

Exclusion Criteria:

For Amputee Subjects:

* Age less than 18 or greater than 75 years
* Unilateral upper limb or multiple limb amputation.
* Amputation due to diabetes or vascular claudication
* No known pending revision surgeries
* Presence of embedded metallic shrapnel or other metal not compatible with MRI scanning
* Presence of traumatic brain injury - permanent or temporary impairments of cognitive, physical, and psychosocial functions with an associated diminished or altered state of consciousness - as indicated by neuropsychological screening, including DVBIC testing, which is currently performed routinely on patients by the TBI program at WRAMC and noted in the patient's medical record
* Known uncontrolled systemic disease- known cancer not in remission
* Known on-going infection
* Lupus
* Kidney disease requiring dialysis, any other systemic disease which might affect ability to participate in this study to its conclusion
* Concurrent participation in another investigational drug or device study for phantom limb pain or participation in the 30 days immediately prior to study enrollment
* Any condition or situation that, in the investigator's opinion, may put the subject at significant risk, confound the study results, or interfere significantly with the subject's participation in the study
* Significant Axis I or II diagnosis determined by a neurologist or psychiatrist in the 6 months prior to entry into the study
* Subjects with lack of effort as determined by the neurologist or physiatrist
* Subjects will be screened for effort using the Test of Memory Malingering (TOMM) first in order to exclude those with blatant exaggeration or malingering

For Control Subjects:

* Age less than 18 or greater than 75 years
* Presence of an amputation
* Presence of embedded metallic shrapnel or other metal not compatible with MRI scanning
* Presence of traumatic brain injury - permanent or temporary impairments of cognitive, physical, and psychosocial functions with an associated diminished or altered state of consciousness - as indicated by neuropsychological screening which is currently performed routinely on patients by the TBI program at WRAMC and noted in the patient's medical record
* Known uncontrolled systemic disease- known cancer not in remission
* Known on-going infection
* Lupus
* Kidney disease requiring dialysis
* Any other systemic disease which might affect ability to participate in this study to its conclusion
* Any condition or situation that, in the investigator's opinion, may put the subject at significant risk, confound the study results, or interfere significantly with the subject's participation in the study
* Significant Axis I or II diagnosis determined by a neurologist or psychiatrist in the 6 months prior to entry into the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2008-02; Primary Completion 2010-02 (Estimated); Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
The identification of brain regions activated before and after treatment with mirror therapy. | 0, 2, and 4 weeks
phantom limb pain as measured using the VAS and McGill | daily for 4 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - National Institutes of Health, Bethesda, Maryland

REFERENCES:
- [Background] Ramachandran VS, Hirstein W. The perception of phantom limbs. The D. O. Hebb lecture. Brain. 1998 Sep;121 ( Pt 9):1603-30. doi: 10.1093/brain/121.9.1603. PMID 9762952
- [Background] Sherman RA, Sherman CJ, Parker L. Chronic phantom and stump pain among American veterans: results of a survey. Pain. 1984 Jan;18(1):83-95. doi: 10.1016/0304-3959(84)90128-3. PMID 6709380
- [Background] Jensen TS, Krebs B, Nielsen J, Rasmussen P. Phantom limb, phantom pain and stump pain in amputees during the first 6 months following limb amputation. Pain. 1983 Nov;17(3):243-256. doi: 10.1016/0304-3959(83)90097-0. PMID 6657285
- [Background] Browder J, Gallagher JP. Dorsal Cordotomy for Painful Phantom Limb. Ann Surg. 1948 Sep;128(3):456-69. doi: 10.1097/00000658-194809000-00011. No abstract available. PMID 17859213
- [Background] Schug SA, Burrell R, Payne J, Tester P. Pre-emptive epidural analgesia may prevent phantom limb pain. Reg Anesth. 1995 May-Jun;20(3):256. No abstract available. PMID 7547671
- [Background] Wall JT. Variable organization in cortical maps of the skin as an indication of the lifelong adaptive capacities of circuits in the mammalian brain. Trends Neurosci. 1988 Dec;11(12):549-57. doi: 10.1016/0166-2236(88)90184-1. No abstract available. PMID 2471312
- [Background] Flor H, Elbert T, Knecht S, Wienbruch C, Pantev C, Birbaumer N, Larbig W, Taub E. Phantom-limb pain as a perceptual correlate of cortical reorganization following arm amputation. Nature. 1995 Jun 8;375(6531):482-4. doi: 10.1038/375482a0. PMID 7777055
- [Background] Grusser SM, Winter C, Muhlnickel W, Denke C, Karl A, Villringer K, Flor H. The relationship of perceptual phenomena and cortical reorganization in upper extremity amputees. Neuroscience. 2001;102(2):263-72. doi: 10.1016/s0306-4522(00)00491-7. PMID 11166112
- [Background] Adrian ED, Zotterman Y. The impulses produced by sensory nerve-endings: Part II. The response of a Single End-Organ. J Physiol. 1926 Apr 23;61(2):151-71. doi: 10.1113/jphysiol.1926.sp002281. No abstract available. PMID 16993780
- [Background] Garraghty PE, Kaas JH. Functional reorganization in adult monkey thalamus after peripheral nerve injury. Neuroreport. 1991 Dec;2(12):747-50. doi: 10.1097/00001756-199112000-00004. PMID 1793816
- [Background] WIESEL TN, HUBEL DH. SINGLE-CELL RESPONSES IN STRIATE CORTEX OF KITTENS DEPRIVED OF VISION IN ONE EYE. J Neurophysiol. 1963 Nov;26:1003-17. doi: 10.1152/jn.1963.26.6.1003. No abstract available. PMID 14084161
- [Background] Elbert T, Flor H, Birbaumer N, Knecht S, Hampson S, Larbig W, Taub E. Extensive reorganization of the somatosensory cortex in adult humans after nervous system injury. Neuroreport. 1994 Dec 20;5(18):2593-7. doi: 10.1097/00001756-199412000-00047. PMID 7696611
- [Background] Lotze M, Laubis-Herrmann U, Topka H, Erb M, Grodd W. Reorganization in the primary motor cortex after spinal cord injury - A functional Magnetic Resonance (fMRI) study. Restor Neurol Neurosci. 1999;14(2-3):183-187. PMID 12671262
- [Background] Merzenich MM, Nelson RJ, Stryker MP, Cynader MS, Schoppmann A, Zook JM. Somatosensory cortical map changes following digit amputation in adult monkeys. J Comp Neurol. 1984 Apr 20;224(4):591-605. doi: 10.1002/cne.902240408. PMID 6725633
- [Background] Pons TP, Garraghty PE, Ommaya AK, Kaas JH, Taub E, Mishkin M. Massive cortical reorganization after sensory deafferentation in adult macaques. Science. 1991 Jun 28;252(5014):1857-60. doi: 10.1126/science.1843843.
- [Background] Ramachandran VS. Blind spots. Sci Am. 1992 May;266(5):86-91. doi: 10.1038/scientificamerican0592-86. No abstract available. PMID 1566041
- [Background] Ramachandran VS, Rogers-Ramachandran D. Synaesthesia in phantom limbs induced with mirrors. Proc Biol Sci. 1996 Apr 22;263(1369):377-86. doi: 10.1098/rspb.1996.0058. PMID 8637922
- [Background] Franz EA, Ramachandran VS. Bimanual coupling in amputees with phantom limbs. Nat Neurosci. 1998 Oct;1(6):443-4. doi: 10.1038/2161. No abstract available. PMID 10196540
- [Background] MacLachlan M, McDonald D, Waloch J. Mirror treatment of lower limb phantom pain: a case study. Disabil Rehabil. 2004 Jul 22-Aug 5;26(14-15):901-4. doi: 10.1080/09638280410001708913. PMID 15497919
- [Background] Lotze M, Flor H, Grodd W, Larbig W, Birbaumer N. Phantom movements and pain. An fMRI study in upper limb amputees. Brain. 2001 Nov;124(Pt 11):2268-77. doi: 10.1093/brain/124.11.2268. PMID 11673327
- [Background] Lotze M, Grodd W, Birbaumer N, Erb M, Huse E, Flor H. Does use of a myoelectric prosthesis prevent cortical reorganization and phantom limb pain? Nat Neurosci. 1999 Jun;2(6):501-2. doi: 10.1038/9145. No abstract available. PMID 10448212
- [Background] Bauer L, O'Bryant SE, Lynch JK, McCaffrey RJ, Fisher JM. Examining the Test Of Memory Malingering Trial 1 and Word Memory Test Immediate Recognition as screening tools for insufficient effort. Assessment. 2007 Sep;14(3):215-22. doi: 10.1177/1073191106297617. PMID 17690378
- [Background] Price DD, Bush FM, Long S, Harkins SW. A comparison of pain measurement characteristics of mechanical visual analogue and simple numerical rating scales. Pain. 1994 Feb;56(2):217-226. doi: 10.1016/0304-3959(94)90097-3. PMID 8008411
- [Background] Melzack R. The short-form McGill Pain Questionnaire. Pain. 1987 Aug;30(2):191-197. doi: 10.1016/0304-3959(87)91074-8. PMID 3670870
- [Background] Buccino G, Binkofski F, Fink GR, Fadiga L, Fogassi L, Gallese V, Seitz RJ, Zilles K, Rizzolatti G, Freund HJ. Action observation activates premotor and parietal areas in a somatotopic manner: an fMRI study. Eur J Neurosci. 2001 Jan;13(2):400-4. PMID 11168545
- [Background] Desmond JE, Glover GH. Estimating sample size in functional MRI (fMRI) neuroimaging studies: statistical power analyses. J Neurosci Methods. 2002 Aug 30;118(2):115-28. doi: 10.1016/s0165-0270(02)00121-8. PMID 12204303
- [Background] Lenth RV. Statistical power calculations. J Anim Sci. 2007 Mar;85(13 Suppl):E24-9. doi: 10.2527/jas.2006-449. Epub 2006 Oct 23. PMID 17060421
- [Derived] Griffin SC, Curran S, Chan AWY, Finn SB, Baker CI, Pasquina PF, Tsao JW. Trajectory of phantom limb pain relief using mirror therapy: Retrospective analysis of two studies. Scand J Pain. 2017 Apr;15:98-103. doi: 10.1016/j.sjpain.2017.01.007. Epub 2017 Mar 7. PMID 28850360